CLINICAL TRIAL: NCT03842449
Title: Impact of Expired Carbon Monoxide Measurement on Smoking Cessation of Pregnant Women - Tobacco Pregnancy Addictive Pregnant Women
Brief Title: Impact of Expired Carbon Monoxide Measurement on Smoking Cessation of Pregnant Women
Acronym: T-CAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 87RC17_0069 (T-CAFE)
Record Dates: First submitted 2019-01-25; First posted 2019-02-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
Keywords: Tobacco; Pregnancy Addictive; Pregnant Women; Stop smoking
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smoking pregnant woman withCO measurement (Experimental)
  Interventions: Diagnostic Test: BabyCO; Other: Biological samples
- Smoking pregnant woman without CO measurement (Other)
  Interventions: Other: Biological samples
- Non Smoking pregnant woman (Other)
  Interventions: Other: Biological samples

INTERVENTIONS:
Diagnostic Test: BabyCO — An expired CO measurement will be performed by BabyCO and the result will be returned to the smoking pregnant woman by the consultant.
  Arms: Smoking pregnant woman withCO measurement
Other: Biological samples — The nature of the samples taken during the delivery are:
  * maternal blood,
  * cord blood
  * placenta fragment

SUMMARY:
France is the country of Europe where the prevalence of pregnant women smokers is the highest (35.9% before pregnancy and in the 3rd quarter 21.8% in 2008).

In the investigator's country, among the smokers of early pregnancy with the usual care, only 30% manage to stop during pregnancy.

Maternal smoking during pregnancy is a clearly identified risk factor for the course of pregnancy and the unborn child.

The measurement of carbon monoxide (CO) expired in pregnancy monitoring consultation is part of the recommendations of the consensus conference "Pregnancy and Tobacco" (ANAES, October 2004) and the parliamentary report on smoking by JL Touraine and D. Jacquat (Feb 2012). However, this recommendation has not entered the current practice. The research aims to justify the clinical relevance of this recommendation by demonstrating the positive impact of expired CO measurement on the rate of discontinuation during pregnancy.

ELIGIBILITY:
Inclusion Criteria :

Group of smoking pregnant women (N = 600):

* Pregnant women declaring themselves smokers (at least one cigarette a day).
* Aged at least 18 years old.
* Consultant at Limoges University Hospital before the 24th week of amenorrhea.
* Desiring to be followed for their entire pregnancy at the Children's.
* Desiring to give birth at the Children's.
* Accepting to participate in the study

Group of strictly non-smoking pregnant women (N = 50):

* Pregnant women :

  * Declaring not to be a smoker (to have been totally weaned for more than one year and to have smoked less than 100 cigarettes in her lifetime) before the beginning of the current pregnancy, and
  * Whose partner and family do not smoke, and
  * Not significantly exposed to tobacco (in their professional environment in particular), and
  * With a CO measurement expired <3 ppm.
* Aged at least 18 years old.
* Consultant at Limoges University Hospital before the 24th SA.
* Desiring to be followed for all their pregnancy and give birth at the Children's Hospital of Limoges.
* Accepting to participate in the study.

Exclusion Criteria :

Group of smoking pregnant women (N = 600) :

* Women with the following social and / or legal criteria: guardianship, curatorship, safeguard of justice.
* Women unable to understand the objectives of the study and the constraints of the protocol.

Group of strictly non-smoking pregnant women (N = 50) :

* Women with the following social and / or legal criteria: guardianship, curatorship, safeguard of justice.
* Women unable to understand the objectives of the study and the constraints of the protocol.
* Women with high blood pressure
* Diabetic woman
* Woman with hypothyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-03-18 (Estimated); Study Completion 2022-03-18 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation on the date of birth | Date of birth
  Evaluate the impact on maternal smoking cessation rate at birth of a strategy combining maternal expired CO measurement, restitution, and outcome comment initiated no later than at the 24th week of amenorrhea and conducted thoughout the whole pregnancy.

SECONDARY OUTCOMES:
Impact on maternal, placental and fetal exposure to the toxic and compounds of tobacco smoke. | Date of birth
  Impact on maternal, placental and fetal exposure to the toxic and compounds of tobacco smoke measured in maternal, cordal blood and placenta by ICP-MS, GC-MS and LC-MS methods
Impact on the intention of breastfeeding on the date of birth | Date of birth
  Impact on the intention of breastfeeding on the date of birth evaluated by a questionnaire
Predictive value of expired CO in relation to maternal-fetal exposure to these toxic and compounds | Date of birth
  Determine the predictive value of expired CO in relation to maternal-fetal exposure to these toxic and compounds
Maternal expired CO on the day of birth | Date of birth
  Maternal expired CO on the day of birth
Determinants of smoking cessation on the day of birth | Date of birth
  Potential determinants of smoking cessation, including: age, parity, precariousness assessed by the EPICES score, history of smoking before pregnancy, expired CO measurement, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No